CLINICAL TRIAL: NCT06740474
Title: A Phase 1a, Blinded, Placebo-Controlled Study of the Safety, Tolerability and Pharmacokinetics of Single- and Multiple-Ascending Doses of ABI-6250 in Healthy Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of ABI-6250 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABI-6250-101
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-02

CONDITIONS: Hepatitis Delta Virus; Hepatitis D
MeSH Terms: conditions — Hepatitis D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part A: SAD Cohorts 1-5, ABI-6250 (Experimental)
- Part A: SAD Cohorts 1-5, Placebo (Placebo Comparator)
- Part A: SAD Food Effect Cohort 6 or 7: ABI-6250 (Experimental)
  Interventions: Drug: ABI-6250
- Part A: SAD Food Effect Cohort 6 (if applicable): Placebo (Placebo Comparator)
- Part B: MAD Cohorts 1-4, ABI-6250 (Experimental)
- Part B: MAD Cohorts 1-4, Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABI-6250 — Single dose (SAD) or once or twice daily dosing over 10 days (MAD)
  Arms: Part A: SAD Food Effect Cohort 6 or 7: ABI-6250
Drug: Placebo — Single dose (SAD) or once or twice daily dosing over 10 days (MAD)
  Arms: Part B: MAD Cohorts 1-4, Placebo

SUMMARY:
This study is designed to assess safety, tolerability, and pharmacokinetics of single ascending doses (SAD) and multiple-ascending doses (MAD) of ABI-6250 in healthy participants. Effect of food will also be evaluated in Part A.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a body mass index (BMI) between ≥18.0 and <32.0 kg/m2 and is in good health (as determined by the Investigator) based on medical history, physical examination, ECG, and clinical laboratory results.
* Female participants must be non-pregnant and have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Day-1 or Day 1 (predose).
* Participants must agree to comply with protocol-specified contraceptive requirements.

Exclusion Criteria:

* Current infection of human immunodeficiency virus (HIV), hepatitis B virus, (HBV), hepatitis C virus (HCV) or acute hepatitis A virus (HAV).
* History of any illness that, in the opinion of the Investigator, might confound the results of the study, pose an additional risk in administering study drug to the subject, or condition known to interfere with the absorption /distribution/ elimination of drugs.
* History of any significant drug-related allergic reactions such as anaphylaxis, Stevens-Johnson Syndrome, urticaria, or multiple drug allergies.
* History of persistent alcohol abuse or illicit drug abuse within 3 years prior to screening.
* Has participated in a clinical study involving administration of either an investigational or a marketed drug within 30 days or 5 half-lives before screening, whatever is longer.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with AEs, premature treatment discontinuation due to AEs and abnormal laboratory results | From enrollment to 10 days after the last dose, at pre-specified timepoints
Area Under the Plasma Concentration Time Curve (AUC) of ABI-6250 | From enrollment to 10 days after the last dose, at pre-specified timepoints
Maximum Observed Plasma Concentration (Cmax) of ABI-6250 | From enrollment to 10 days after the last dose, at pre-specified timepoints
Time to Cmax (Tmax) of ABI-6250 | From enrollment to 10 days after the last dose, at pre-specified timepoints
Apparent Terminal Elimination Half Life (t 1/2) of ABI-6250 | From enrollment to 10 days after the last dose, at pre-specified timepoints
Apparent Systemic Clearance (CL/F) of ABI-6250 | From enrollment to 10 days after the last dose, at pre-specified timepoints
Apparent Volume of Distribution (Vz/F) of ABI-6250 | From enrollment to 10 days after the last dose, at pre-specified timepoints
Dose normalized AUCs and Cmax of ABI-6250 | From enrollment to 10 days after the last dose, at pre-specified timepoints

SECONDARY OUTCOMES:
Comparison of plasma AUC between fasted and fed treatments | From enrollment to 10 days after the last dose, at pre-specified timepoints
Comparison of AUC between fasted and fed treatments | From enrollment to 10 days after the last dose, at pre-specified timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- New Zealand Clinical Research, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No